CLINICAL TRIAL: NCT01332084
Title: Assessment of the Feasibility of a SOTI With Hypoallergenic (H.A.) Cereals in Children With Diagnosed IgE-mediated Allergy to Wheat
Brief Title: Use of Hypoallergenic (H.A.) Cereals in Children With Diagnosed Allergy to Wheat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.19.INF
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Food Allergy
Keywords: SOTI; tolerance; desensitization; challenge test; HA wheat cereals
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypoallergenic wheat cereals (Experimental): HA wheat cereal used in a SOTI test
  Interventions: Other: HA wheat cereals

INTERVENTIONS:
Other: HA wheat cereals — HA wheat cereals used in SOTI test and as part of desensitization plan

SUMMARY:
The investigators plan to launch a Specific Oral Tolerance Induction (SOTI) pilot study in order to assess the efficacy and the safety of hypoallergenic (H.A.) wheat cereals, for children with allergy to wheat. The study has the potential to offer a desensitization treatment option for children allergic to wheat.

The investigators hypothesize that H.A. wheat cereals have similar efficacy with less side effects than native wheat cereals.

DETAILED DESCRIPTION:
In this pilot study, the investigators aim to assess the feasibility of a SOTI (Specific Oral Tolerance Induction) with hypoallergenic (H.A.) cereals in children with diagnosed IgE-Mediated allergy to wheat.

This is a multi centre, open, pilot study testing 1 product.10 children of any ethnicity aged from 1 to 12 years old with diagnosed allergy to wheat will be eligible to participate in the study. The duration of the treatment will be 6 months with a minimum of 1 month of daily consumption of the hydrolyzed wheat cereals.

Each subject will feed with a quantity of the assigned study product according to the SOTI. The SOTI will be performed at the hospital under the control of qualified doctors and nurses.

The study product is administered starting with very low dosages, which are increased stepwise every 30 minutes up to an amount equivalent to the usual daily oral intake. Thereafter, the study product corresponding to the maximum dose tolerated is given in a maintenance dose in one serve every day until the final visit during which a challenge test with wheat will be performed to assess the tolerance of whole wheat.

ELIGIBILITY:
Inclusion Criteria:

* Infant of any ethnicity aged between 1 to 12 years old at the time of enrollment and
* Positive Skin Prick Test (SPT) to wheat and/or Positive specific IgE to wheat and
* Immediate positive reaction (IgE-type reaction) to wheat as shown by provocation test done a maximum 1 year before the enrollment to the study or an unambiguous history for wheat allergy as evaluated by the investigator and
* Having obtained his/her signed legal representative's informed consent

Exclusion Criteria:

* Child on systemic drugs (potentially affecting the allergic reactions e.g. antihistamines) according to half-life at time of enrollment or
* Congenital illness or malformation that may affect normal growth (especially immunodeficiency) or
* Child with uncontrolled asthma or
* Child whose parents/caregivers cannot be expected to comply with treatment or
* Child currently participating in another interventional clinical trial.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Specific Oral Tolerance Induction (SOTI) with hypoallergenic wheat in children allergic to wheat | 6 months
  The primary outcome is to document Clinical examination for presence or absence of immediate adverse reaction during the SOTI with evaluation of the maximum dose tolerated during the SOTI.
  Symptoms related to allergic reactions during the SOTI (if applicable)will be recorded in the CRF.

SECONDARY OUTCOMES:
assess allergic reactions to a challenge test to wheat | 6 months
  challenge test will be performed at the end of the treatment with HA cereals. Other blood immunological parameters will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Lauener, Prof MD, Principal Investigator — Universitäts-Kinderklinik Zürich; Jacqueline Wassenberg, MD, Principal Investigator — Département médico-chirurgical de pédiatrie, CHUV, Lausanne; Philippe Eigenmann, MD, Principal Investigator — Adult&Child Allergy Unit, Geneva
Locations (2):
- Switzerland (2):
  - Adult&Child Allergy Unit, HUG, Geneva
  - Unité d'immunologie, allergologie et rhumatologie pédiatrique Département médico-chirurgical de pédiatrie CHUV, Lausanne